CLINICAL TRIAL: NCT01851135
Title: Neuropsychological Impairment and Quality of Life in Neurofibromatosis Type 1
Acronym: NF1-QDV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Université d'Angers (Angers, France) (Unknown); Association Neurofibromatoses et Recklinghaüsen (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: RC12_0130
Record Dates: First submitted 2013-04-24; First posted 2013-05-10 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Neurofibromatosis Type 1
Keywords: Quality of life; Neuropsychological disorders; Neurofibromatosis type 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with NF1 (Experimental)
  Interventions: Other: Neuropsychological examination and quality of life measures
- Healthy controls (Other)
  Interventions: Other: Neuropsychological examination and quality of life measures

INTERVENTIONS:
Other: Neuropsychological examination and quality of life measures

SUMMARY:
The main objective of the study is to investigate the determinants of the quality of life in children and adults with Neurofibromatosis type 1 (NF1) and more particularly the specific impact of neuropsychological deficits. In fact, cognitive impairment is currently considered as one of the most pervasive features of this genetic disorder but its relationship with the worsening of quality of life found in this population has not been directly investigated to date.

Secondary objectives of this study are (i) to compare neuropsychological and quality of life measures between patients and healthy controls matched by age, gender and education level, (ii) to contrast neuropsychological deficits incidence between patients and controls, and (iii) to differentiate NF1 children's self versus hetero-assessment of quality of life.

The main hypothesis of this study is that the neuropsychological impairment classically identified in this clinical population will be associated to the quality of life's worsening both in children and adults.

DETAILED DESCRIPTION:
The study cohort will consist of 150 patients with NF1 (100 adults and 50 children) recruited from the Neurofibromatosis Clinic at the University Hospital in Nantes and Créteil (France). A sample of 150 healthy controls (100 adults and 50 children) will also be recruited from sport and leisure clubs to serve as a normally developing control group.

The protocol assessment includes a standard and thorough neuropsychological examination specific to children and adults, to investigate the different aspects of cognitive domains: language, visuoperceptive and visuomotor abilities, memory, attention, executive function and intelligence skills. Quality of life is measured by a questionnaire specifically adapted to children and adults.

Other factors linked to the NF1 disease (familial or sporadic form, severity and visibility) and to demographic characteristics (sex, age, education level) will be taken into account to study their respective impact on quality of life, as compared with neuropsychological measures.

ELIGIBILITY:
Inclusion Criteria for Patients :

* NF1 diagnosis following National Institutes of Health criteria (1988)
* Age: 8-12 years for children, 18-59 years for adults
* Signed informed written consent (parent and patient for children, patient for adults)
* French speaking
* Resident in France

Inclusion Criteria for Healthy controls:

* Absence of NF1 diagnosis, learning disabilities, intellectual precocity
* Age: 8-12 years for children, 18-59 years for adults
* Signed informed written consent (parent and healthy control for children, healthy control for adults)
* French speaking
* Resident in France

Exclusion Criteria:

* Uncorrectable hearing of visual impairment
* History of psychiatric illness
* Neuropsychological investigation in the last 6 months
* Insufficient language usage
* Any other known history of central nervous system pathology or neuropathological complications of NF1

Ages: 8 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 286 (Actual)
Dates: Start 2013-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Quality of life as measured by the questionnaires used in children and adults | at day 0 for adults; at 4 weeks for children
  Several domains in relation with quality of life (self perception, well-being, social life, emotions, etc.)

SECONDARY OUTCOMES:
Scores obtained from neuropsychological tests (composite measure) | at day 0 and 2 weeks for adults; at day 0, 2 weeks and 4 weeks for children
  The neuropsychological tests used in this study evaluate different domains: language, visuoperceptive and visuomotor abilities, memory, attention, executive function and intelligence skills.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Barbarot, MD, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - Assistance Publique - Hôpitaux de Paris (Hôpital Henri Mondor), Créteil
  - Centre Hospitalier Universitaire de Nantes, Nantes